CLINICAL TRIAL: NCT00887068
Title: Randomized Controlled Study of Post-transplant Azacitidine for Prevention of Acute Myelogenous Leukemia and Myelodysplastic Syndrome Relapse (VZ-AML-PI-0129)
Brief Title: Controlled Study of Post-transplant Azacitidine for Prevention of Acute Myelogenous Leukemia and Myelodysplastic Syndrome Relapse (VZ-AML-PI-0129)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0503; NCI-2012-01259 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Leukemia; AML; MDS
Keywords: Leukemia; Acute myelogenous leukemia; AML; Myelodysplastic syndrome; MDS; Remission; Allogeneic stem cell transplant; Allotx; Azacitidine; 5-Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacitidine (Experimental): Azacitidine 32 mg/m^2 given through a needle under the skin for five consecutive days of each 28 day cycle and the maximum treatment will be 12 cycles.
  Interventions: Drug: Azacitidine
- No Azacitidine (No Intervention): Standard treatment post allogeneic transplant is supportive care only.

INTERVENTIONS:
Drug: Azacitidine — 32 mg/m^2 given through a needle under the skin for five consecutive days of each 28 day cycle and the maximum treatment will be 12 cycles.
  Other Names: 5-Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Azacitidine

SUMMARY:
The goal of this clinical research study is to learn if Vidaza (azacitidine) will help to control the disease in patients with AML, CMML, or MDS after an allogeneic (donor) stem cell transplant. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Azacitidine is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in a flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive azacitidine.
* If you are in Group 2, you will not receive azacitidine.

Study Drug Administration:

If you are in Group 1, you will receive azacitidine through a needle under your skin on Days 1-5 of each cycle.

Each cycle is 28 days long.

Your dose of azacitidine may be lowered or stopped if certain side effects develop.

Study Visits:

About 2 or 3 days before each cycle and, if your doctor thinks it is needed, on Day 3 of each cycle and 1 time during Weeks 2 and 3 of each cycle, blood (about 4 teaspoons each time) will be drawn for routine tests.

At 3, 6, and 12 months after the stem cell transplant:

* You will have a complete medical history and physical exam.
* Blood (about 4 teaspoons each time) will be drawn for routine tests.
* You will have a bone marrow aspiration to check the status of the disease.

You may come back for study visits more often if the doctor thinks it is needed.

While on study, you will need to stay in Houston for about 3 months after the transplant (this is standard after stem cell transplants).

Length of Study:

You will be on study treatment for up to 1 year (up to 12 cycles of azacitidine). You will be taken off study early if you experience intolerable side effects or the disease gets worse.

End-of-Treatment Visit:

After you complete the planned treatment with azacitidine, you will have an end-of-treatment visit:

* You will have a complete medical history and physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspiration to check the status of the disease.

This is an investigational study. Azacitidine is FDA approved and is commercially available for the treatment of myelodysplastic syndrome.

Up to 246 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of AML (World Health Organization classification: >=20% blasts in the bone marrow and / or peripheral blood) or MDS (International Prognostic Scoring System intermediate-1 or higher) that at the time of allogeneic transplantation were in: - Induction Failure, relapsed disease or second or greater remission; patients in first complete remission that required more than 1 cycle of treatment to achieve the remission, or that have AML evolving from MDS, or that had the following abnormalities: FLT3 mutation, deletion of chromosome 5 or 7, MLL gene rearrangement, or more than or equal to 3 cytogenetics abnormalities. Patients with de novo or therapy-related MDS, CMML, or AML are also eligible, regardless of cytogenetics or molecular rearrangements.
2. Biphenotypic Leukemia that at the time of allogeneic transplantation was in induction failure, relapsed disease, first, second or greater remission.
3. Patients must be in complete remission post transplant.
4. Patient may be enrolled 40 to 100 days after transplant.
5. Age 18 to 75 years old.
6. Serum creatinine < 1.8 mg/dL or creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault Equation*. a. Males(mL/min):(140-age)*IBW(kg) / 72*(serum creatinine(mg/dl)) b. Females(mL/min):0.85*(140-age)*IBW(kg) / 72*(serum creatinine(mg/dl)).
7. Serum direct bilirubin < 1.5 mg/dL (unless Gilbert's syndrome).
8. SGPT </= 200 IU/ml unless related to patient's malignancy.
9. Be able to understand and sign informed consent.

Exclusion Criteria:

1. Active uncontrolled infection.
2. Presence of uncontrolled graft-versus-host disease.
3. Patients that underwent allogeneic transplantation as a treatment of graft failure.
4. Pregnancy or breast-feeding (women of childbearing potential, any female who has experienced menarche and who has not undergone surgical sterilization or is not post-menopausal with a positive serum pregnancy test.
5. Known or suspected hypersensitivity to azacitidine or mannitol.
6. Patients with advanced malignant hepatic tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2009-04-21 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Oran B, de Lima M, Garcia-Manero G, Thall PF, Lin R, Popat U, Alousi AM, Hosing C, Giralt S, Rondon G, Woodworth G, Champlin RE. A phase 3 randomized study of 5-azacitidine maintenance vs observation after transplant in high-risk AML and MDS patients. Blood Adv. 2020 Nov 10;4(21):5580-5588. doi: 10.1182/bloodadvances.2020002544. PMID 33170934
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from September 2009 to April 2017 for high risk subjects with acute myelogenous leukemia (AML) and myelodysplastic (MDS) patients who have undergone an allogeneic transplant.
Pre-assignment Details: Patients were randomized to receive azacitidine (AZA) or standard of care 40 to 100 days after allo SCT.
Groups:
- AZA Group: Subjects randomized to the AZA treatment will receive 32 mg/m2 for 5 consecutive days of each 28 day cycle and the maximum treatment will be 12 cycles. Each cycle will consist of approximately 28 days, allowing the possibility that treatment within a cycle may be delayed for up to 4 weeks due to organ toxicity or hematologic toxicity.
- Standard of Care Group: Best standard of care (ie, no maintenance)
Period: Overall Study
Arm/Group | AZA Group | Standard of Care Group
Started | 93 | 94
Completed | 87 | 94
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Didn't meet eligibility to start cycle 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled patients were randomly assigned; in a 1:1 ratio; to 12 cycles of azacitidine (at a dose of 32 mg per square meter of body surface area per day, administered by subcutaneous injections for 5 days every 4 weeks) or to observation (no further treatment). The randomization was stratified by disease (AML, MDS, biphenotypic leukemia).
Groups:
- Total: Total of all reporting groups
Arm/Group | AZA Group | Standard of Care Group | Total
Number analyzed (Participants) | 87 | 94 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 73 | 144
  >=65 years | 16 | 21 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 51 | 57 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 79 | 92 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 87 | 94 | 181
Disease Strata [Count of Participants; unit: Participants] — The randomization was stratified by disease (AML, MDS, biphenotypic leukemia).
  Participants
    AML | 67 | 67 | 134
    MDS | 26 | 26 | 52
    Biphenotypic Leukemia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS)
Description: The time that a participant survives without relapse of the disease.
Time Frame: 3 years
Measure: Median (Standard Deviation); unit: years
Arm/Group | AZA Group | Standard of Care Group
Number analyzed (Participants) | 87 | 94
years | 2.1 (.43) | 1.3 (.43)

2. Secondary Outcome: Overall Survival (OS)
Time Frame: 3 years
Measure: Median (Standard Deviation); unit: years
Arm/Group | AZA Group | Standard of Care Group
Number analyzed (Participants) | 87 | 94
years | 2.5 (.85) | 2.6 (.85)

ADVERSE EVENTS:
Time Frame: From time of enrollment dependent on randomization would be one month from last day of study drug or one year if in standard of care group.
Arm/Group | AZA Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/87 | 1/94
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/94
Other Adverse Events (participants affected / at risk) | 29/87 | 19/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZA Group (N=87) | Standard of Care Group (N=94)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 | 1
Poor Graft function (Blood and lymphatic system disorders) | 29 | 2
Infection (Infections and infestations) | 0 | 19
Gastrointestetinal (Gastrointestinal disorders) | 0 | 12
Hepatic (Hepatobiliary disorders) | 8 | 5
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Skin (Skin and subcutaneous tissue disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT00887068/Prot_SAP_000.pdf